CLINICAL TRIAL: NCT06097598
Title: Prevalence of Irritable Bowel Syndrome in Medical Students in the Middle East and North Africa
Brief Title: Prevalence of Irritable Bowel Syndrome in Medical Students Africa
Acronym: Irritablebowel
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: AsyutUniversity (Unknown)
Responsible Party: Principal Investigator, Zeinab Galal Eldeen Abdelhamid, Demonstrator, Assiut University
Other Study IDs: Irritable
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Faculty of Medicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study was to assess the prevalence of IBS among medical students in the Middle East and North Africa and to investigate the sociodemographic, lifestyle, and clinical factors associated with IBS. A better understanding of IBS correlates is expected to improve our therapeutic approach to IBS in this population.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a multifactorial chronic disease characterized with functional gastrointestinal disorder which affects the quality of life of the patient. Until now the pathophysiology of IBS was not completely understood but it has been related to multiple mechanisms like: visceral hypersensitivity, Brain-gut axis, post infectious inflammation and genetic abnormalities.(1) Many demographic and environmental factors are considered risk factors for the condition like: sex, age, BMI, social status and life style(2). IBS outspreaded all over the world varying between 14.7% to 16.5% in east Asian countries(3,4). As IBS is diagnosed mainly clinically, many scales have been developed to provide the best sensitivity for diagnosing the condition. The recent common criteria for diagnosing are ROME III and ROME VI. A meta-analysis conducted by Oka et al the pooled prevalence of IBS in 53 surveys that used the Rome III criteria from 38 countries was 9.2% (95% CI 7.6-10.8; I2 = 99.7%). Contrary, the pooled IBS prevalence among the 6 surveys that used the Rome IV criteria from 34 countries was 3.8% (95% CI 3.1-4.5; I2 = 96.6%)(5). The different prevalence rates are probably justified by the multifactorial nature of the disease and the various social status and environments from a country to another. However, there wasn't enough studies could define the prevalence of IBS among middle-eastern countries. The prevalence of IBS varies depending on socioeconomic factors, sex, and age. University students in the Middle East and North Africa are affected by many Lifestyle factors that participate in IBS by one way or another such as unhealthy eating habits (junk or fast food), cigarette smoking, physical inactivity and the fact that they're living low-income countries. IBS has also been associated with psychological factors such as stress, depression, and anxiety. Additionally, as their young age genetic factors and positive family history are implicated. Medical students, are more likely exposed to IBS risk factors as they have limited access to healthy meals, financial constraints, and a excessive exposure to stress secondary to their exceedingly demanding education and frequent examinations. Thus, they are more probably to develop IBS than other population subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Medical students enrolled in from medical schools located in the Middle East and North Africa.

Exclusion Criteria:

* 1- History of significant comorbidities 2- Participants with definite or suspected history of inflammatory bowel disease, celiac disease, Lactose intolerance or peptic ulcer disease. 3- Psychiatric patients or patients on antidepressant treatment or using psychotropic drugs affecting their cognitive ability.

Max Age: 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Medical students enrolled in from medical schools located in the Middle East and North Africa.
Sampling Method: Non-Probability Sample
Enrollment: 1131 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Describe the prevalence of IBS among medical students | 6 month
  assess the prevalence of IBS among medical students in the Middle East and North Africa and to investigate the sociodemographic,
  Page 3 of
  lifestyle, and clinical factors associated with IBS. A better understanding of IBS correlates is expected to improve our therapeutic approach to IBS in this population.

REFERENCES:
- [Background] Camilleri M. Peripheral mechanisms in irritable bowel syndrome. N Engl J Med. 2012 Oct 25;367(17):1626-35. doi: 10.1056/NEJMra1207068. No abstract available. PMID 23094724
- [Background] Black CJ, Ford AC. Global burden of irritable bowel syndrome: trends, predictions and risk factors. Nat Rev Gastroenterol Hepatol. 2020 Aug;17(8):473-486. doi: 10.1038/s41575-020-0286-8. Epub 2020 Apr 15. PMID 32296140
- [Background] Seger S, Nasharuddin NNB, Fernandez SL, Yunus SRBM, Shun NTM, Agarwal P, Burud I. Prevalence and factors associated with irritable bowel syndrome among medical students in a Malaysian private university: a cross sectional study. Pan Afr Med J. 2020 Oct 13;37:151. doi: 10.11604/pamj.2020.37.151.21716. eCollection 2020. PMID 33425184
- [Background] Basandra S, Bajaj D. Epidemiology of Dyspepsia and Irritable Bowel Syndrome (IBS) in Medical Students of Northern India. J Clin Diagn Res. 2014 Dec;8(12):JC13-6. doi: 10.7860/JCDR/2014/10710.5318. Epub 2014 Dec 5. PMID 25653974
- [Background] Oka P, Parr H, Barberio B, Black CJ, Savarino EV, Ford AC. Global prevalence of irritable bowel syndrome according to Rome III or IV criteria: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2020 Oct;5(10):908-917. doi: 10.1016/S2468-1253(20)30217-X. Epub 2020 Jul 20. PMID 32702295